CLINICAL TRIAL: NCT01172431
Title: A Comparison of Indapamide SR 1.5 mg With Hydrochlorothiazide 25 mg, in Combination With an ACE-inhibitor, in Old Patients With Mild to Moderate Renal Insufficiency and Hypertension
Brief Title: Indapamide Versus Hydrochlorothiazide in Elderly Hypertensive Patients With Renal Insufficiency
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Xiaoping Chen, Xiaoping Chen, professor, West China Hospital of Sichuan University., West China Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WestChinaH
Record Dates: First submitted 2010-07-26; First posted 2010-07-29 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2014-06

CONDITIONS: Hypertension; Renal Insufficiency
Keywords: hypertension; renal insufficiency; indapamide; hydrochlorothiazide
MeSH Terms: conditions — Hypertension; Renal Insufficiency | interventions — Indapamide; Hydrochlorothiazide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Indapamide (Experimental): Indapamide SR 1.5mg qd
  Interventions: Drug: Indapamide
- Hydrochlorothiazide (Active Comparator): Hydrochlorothiazide 25mg qd
  Interventions: Drug: Hydrochlorothiazide

INTERVENTIONS:
Drug: Indapamide — Indapamide SR 1.5mg qd
  Arms: Indapamide
Drug: Hydrochlorothiazide — Hydrochlorothiazide 25mg qd
  Arms: Hydrochlorothiazide

SUMMARY:
The purpose of this study is to evaluate the effects of indapamide SR 1.5 mg on renal function, endothelial function, blood pressure variability by comparison with hydrochlorothiazide 25 mg, in patients with Mild to Moderate Renal Insufficiency and Hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Creatinine clearance 30 to 90 mL/min/1.73 m2, with variations of less than 20 percent in the 2 weeks before the screening evaluation.
* Diagnosed hypertension according to guidelines or having taken anti-hypertension drugs.
* Aged between 65 and 85 years.
* Willingness to provide written, informed consent.
* Ability to adhere to study protocol.

Exclusion Criteria:

* Secondary hypertension.
* Diabetes mellitus.
* Atrial flutter/atrial fibrillation.
* Symptoms of congestive heart failure (NYHA III-IV) or there is evidence that left ventricular EF < 40%.
* Recent (< 6 months) myocardial infarction or cerebrovascular ischemic symptoms.
* Recent (< 3 months) or planned coronary revascularization: PCI (percutaneous coronary intervention)/CABG (coronary artery by-pass graft).
* Severe valvular heart disease.
* History of hypersensitivity to indapamide, thiazides or to any of the components of the products.
* Any current condition or other disease known to interfere significantly with the absorption, distribution, metabolism or excretion of study drugs.
* Participation to another investigational study in the last 3 months.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 240 (Actual)
Dates: Start 2010-09; Primary Completion 2012-03 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
renal function | 1 year
  Effects of indapamide SR 1.5 mg on renal function by comparison with hydrochlorothiazide 25 mg, in patients with Mild to Moderate Renal Insufficiency and Hypertension.

SECONDARY OUTCOMES:
endothelial function | 1 year
  Effects of indapamide SR 1.5 mg on endothelial function by comparison with hydrochlorothiazide 25 mg, in patients with Mild to Moderate Renal Insufficiency and Hypertension.
blood pressure variability | 1 year
  Effects of indapamide SR 1.5 mg on blood pressure variability by comparison with hydrochlorothiazide 25 mg, in patients with Mild to Moderate Renal Insufficiency and Hypertension

CONTACTS AND LOCATIONS:
Overall Officials: Xiao P Chen, master, Principal Investigator — West China Hospital
Locations (1):
- Department of Cardiology, West China Hospital, Sichuan University, Chengdu, Sichuan, China